CLINICAL TRIAL: NCT06426615
Title: Connectivity and Neural Signatures of Consciousness In Unresponsive States (CONSCIUS) - a Study of Brain Activity in Disorders of Consciousness
Brief Title: Connectivity and Neural Signatures of Consciousness in Unresponsive States
Acronym: CONSCIUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: s67062
Record Dates: First submitted 2024-03-29; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-03

CONDITIONS: Acute Brain Injury; Traumatic Brain Injury; Consciousness Disorders; Seizures
Keywords: Consciousness; Seizures; Neural dynamics; Intracranial recordings and stimulation
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic; Consciousness Disorders; Seizures

STUDY DESIGN:
Intervention Model Description: Prospective inclusion of patients implanted with intracranial electrodes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute brain injury (Experimental): Patients with acute brain injury with reduced consciousness that undergo multimodal intracranial monitoring, or with suspected seizures
  Interventions: Device: Intracranial electrodes

INTERVENTIONS:
Device: Intracranial electrodes — Placement of intracranial electrodes in the cortico-subcortical system
  Other Names: Depth electrodes

SUMMARY:
The CONSCIUS study is a prospective, interventional study including patients with acute brain injury and impaired consciousness implanted with intracranial electrodes. The aim of the study is to investigate seizures and thalamocortical neural dynamics underlying behavioral unresponsiveness.

DETAILED DESCRIPTION:
Individuals with severe brain injury often require extensive treatment in intensive care units (ICU) and hospitalization wards while uncertainty prevails about the recovery of consciousness and cognitive abilities. Especially in the acute phase after injury, treatment decisions have a tremendous impact on outcome, but rely on assessments of behavioral responsiveness which are known to be unreliable and subject to many confounders. Objective, quantifiable diagnostic and prognostic measures that can be deployed at the bedside during the ICU stay are lacking. Development of new metrics are hampered by our lack of a fundamental understanding of (i) thalamocortical network mechanisms underlying consciousness and (ii) brain-injury induced neural dynamics impacting both consciousness and outcome. Continuous EEG monitoring has been used to aid in this respect to (i) predict recovery of consciousness and outcome, and (ii) diagnose nonconvulsive seizures in unresponsive patients. Although promising, it lacks sensitivity, spatial resolution, and causal power. There is an urgent need for techniques allowing high-precision detection of pathological dynamics, patient stratification and prediction of a capacity for consciousness recovery in acute unresponsive patients with brain injury. Intracranial electrodes as part of multimodal monitoring in subjects with impaired consciousness and severe brain injury allow continuous bedside recordings of high spatiotemporal resolution in different network nodes and allows inducing brain perturbations, transcending correlational evidence of network analysis. This technique could increase the detection and treatment of nonconvulsive seizures contributing to brain injury and unresponsiveness and simultaneously allows to study networks supporting consciousness. This can lead to new diagnostic and prognostic biomarkers for recovery based on thalamocortical profiles of activity, reactivity (complexity) and connectivity, ultimately paving to way for the development of biomarker-driven treatments to support early recovery such as deep brain stimulation. Eventually this can contribute to clinical decision making: abstaining from aggressive treatment in patients with no potential for recovery, and more importantly, continuing treatment in subjects with a responsive brain but without clear behavioural correlate.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Brain injury of any kind, with impaired consciousness or suspected seizures

Exclusion Criteria:

* < 18 years old
* Known pregnancy
* Any condition that, in the judgement of the investigator, makes participation in the study unsafe or unfeasible (e.g., irreversible coagulopathy, large intracranial tumors, surgical technical problems…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of electrographic epileptiform activity (ictal and ictal-interictal continuum activity) on intracranial versus scalp electroencephalography (EEG). | A maximum of 4 weeks after electrode implantation.
  The primary aim is to compare the incidence of ictal and ictal-interictal continuum epileptiform activity on intracranial versus scalp EEG.

SECONDARY OUTCOMES:
Correlating neural activity patterns (local field potentials and complexity) with behavioral responsiveness (measured using the Coma Recovery Scale-Revised). | A maximum of 4 weeks after electrode implantation.
  Correlation of profiles of neural activity and reactivity with the behavioral state using the Coma Recovery Scale-Revised (CRS-R).
Acute effects of electrical stimulation on behavioral responsiveness (measured using the Coma Recovery Scale-Revised). | During electrical stimulation trials, performed in the first 4 weeks after electrode implantation.
  Effects of electrical stimulation on behavioral responsiveness will be measured using the Coma Recovery Scale Revised (CRS-R).
Correlation of neural activity profiles with long-term outcome (Coma Recovery Scale-Revised and Glasgow Outcome Scale-Extended) | At 6 months and 1 year follow-up.
  Profiles of activity and reactivity identified during the acute stage of the disease will be correlated with long-term outcome measures mainly at 6m and 1y, using Coma Recovery Scale-Revised and Glasgow Outcome Scale-Extended.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Theys, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZLeuven, Leuven, Vlaams-Brabant, Belgium